CLINICAL TRIAL: NCT00629434
Title: A Comparison of Diabetes Group Education as Administered Through Telemedicine Versus as Administered in Person
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: State University of New York - Upstate Medical University (Other)
Responsible Party: Roberto Izquierdo, MD, SUNY Upstate Medical University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UMU IRB # 4510F; UMU IRB # 4510F
Record Dates: First submitted 2008-02-25; First posted 2008-03-06 (Estimated); Last update posted 2021-10-06 (Actual); Status verified 2021-10

CONDITIONS: Diabetes Mellitus
Keywords: Diabetes Education; Telemedicine
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): This arm will receive diabetes education via telemedicine
  Interventions: Other: diabetes education via telemedicine
- 2 (Active Comparator): diabetes education in-person
  Interventions: Other: diabetes education in-person

INTERVENTIONS:
Other: diabetes education via telemedicine — This arm will receive diabetes group education via telemedicine
  Arms: 1
Other: diabetes education in-person — In this arm the group of patients with diabetes will receive diabetes education in-person
  Arms: 2

SUMMARY:
This study compares group diabetes education in-person versus via telemedicine

DETAILED DESCRIPTION:
Diabetes education is important in the treatment of the person with diabetes. A diabetes self-management education program not only educates the patient and his/her family to the basics of diabetes care but also integrates diabetes care into daily life while providing coping skills to adjust to this chronic illness. Unfortunately, comprehensive diabetes care is not available to all persons with diabetes. One obstacle to the provision of comprehensive diabetes care is the unavailability of a diabetes treatment center. many people with diabetes live too far or do not have the transportation to be able to attend education programs that met national standards. We have shown that telemedicine is an effective means to provide comprehensive 1:1 individualized diabetes education to persons with diabetes. We now propose to test the hypothesis that diabetes groups education classes can be provided effectively through telemedicine technology to individuals living in rural areas. Patients with diabetes will received diabetes education via teleconferencing from our Joslin Diabetes center. The participants will be assessed before and after diabetes education via telemedicine using measures of glycemia (A1c) and assessments of patient satisfaction, emotional well being, and behavioral change and compared to results from participants attending our diabetes education classes in-person.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 or type 2 diabetes mellitus
* age > 18 years

Exclusion Criteria:

* Profound vision loss
* Severe hearing impairment

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2001-06; Primary Completion 2008-06 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
A1c | baseline, 3 mo post intervention, 6 mo post intervention

SECONDARY OUTCOMES:
PAID scale | baseline, 3 and 6 months post intervention
Diabetes Treatment Satisfaction Questionnaire | Baseline, 3 and 6 months post intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Joslin Diabetes Center Affiliate at SUNY Upstate Medical University, Syracuse, New York, United States